CLINICAL TRIAL: NCT06610383
Title: Effect of Circadian Rhythm of Adrenal Glucocorticoid on Pain, Swelling, and Trismus After Surgical Removal of Mandibular Third Molars
Brief Title: Evaluation of the Effect of Circadian Rhythm of Adrenal Glucocorticoids After Third Molar Extraction
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Muhammet Yasin Pektaş, Research Asistant, Afyonkarahisar Health Sciences University
Other Study IDs: 21.KARİYER.008
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Wisdom Teeth
Keywords: wisdom teeth; circadian rhythm; steroid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 (08:30 group (n=20)): Patients in this group will spit into 1.5 ml tubes at 08:30 in the morning before starting the impacted tooth surgery and 48 hours after the surgery, and these tubes will be stored in the refrigerator at -22 degrees. The samples in these tubes will then be examined with ELISA kits and the numerical data of adrenal glucocorticoids in the saliva will be obtained. The patients will fill out the Visual Analog Scale and OHIP-14 forms a total of five times: 6 hours, 24 hours, 48 hours, 72 hours and 7 days after the surgery.
  Interventions: Procedure: Surgical extraction of wisdom teeth in the morning
- Group 2 (15:30 group (n=20)): Patients in this group will spit into 1.5 ml tubes at 15:30 in the morning before starting the impacted tooth surgery and 48 hours after the surgery, and these tubes will be stored in the refrigerator at -22 degrees. The samples in these tubes will then be examined with ELISA kits and the numerical data of adrenal glucocorticoids in the saliva will be obtained. The patients will fill out the Visual Analog Scale and OHIP-14 forms a total of five times: 6 hours, 24 hours, 48 hours, 72 hours and 7 days after the surgery.
  Interventions: Procedure: Surgical extraction of wisdom teeth in the afternoon

INTERVENTIONS:
Procedure: Surgical extraction of wisdom teeth in the morning — The patients in this group underwent impacted tooth surgery at 08:30 in the morning.
  Groups: Group 1 (08:30 group (n=20))
Procedure: Surgical extraction of wisdom teeth in the afternoon — Impacted tooth surgery was performed on the patients in this group at 15:30.
  Groups: Group 2 (15:30 group (n=20))

SUMMARY:
This study aimed to investigate the effects of wisdom tooth surgery performed at different times of the day on pain, swelling and trismus based on changes in the circadian rhythm in the adrenal glands in patients aged between 18-25 years who applied to the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Afyonkarahisar Health Sciences University with complaints of pain and swelling due to wisdom teeth.

DETAILED DESCRIPTION:
This clinical study was conducted on 20 patients who applied to the Afyonkarahisar Health Sciences University (AFSU) Faculty of Dentistry, Department of Oral and Maxillofacial Surgery between November 2021 and July 2022 for surgical extraction of mandibular impacted third molars in the same impaction class (Mesioangular-Pell and Gregory class II-B) bilaterally. This study was created by including 20 patients who applied to the AFSÜ Faculty of Dentistry, Oral, Dental and Maxillofacial Surgery Clinic due to the presence of impacted teeth and/or complaints caused by their impacted teeth, and who were decided to have symmetrical, bilateral, bone-retained (Mesioangular) third molars in the mandible extracted as a result of clinical examination and radiographic evaluations.

Participation in this study was completely up to the participant. If the participant did not want to participate in the study or withdrew, the doctor still applied the most appropriate treatment plan for the participant.

During the surgery for your wisdom teeth, we took a saliva sample from the participant before anesthesia, on the 2nd and 7th postoperative days, and measured the amount of steroids secreted from your body through your saliva. The participant's pain, swelling, and trismus values were assessed using reference points on your face and pain scales on the day he/she came to the surgery, the 2nd day, and the 7th day. The study has no risks or discomfort. Based on the results of this study, surgeons will be able to evaluate the effects of adrenal steroids at different times of the day and determine when their procedures will be more comfortable. Participants did not incur any financial burden by participating in the study, and no payment was made to the participants. The researchers will use the participants' personal information to conduct the study and statistical analyses, but the participants' identities will be kept confidential. Ethics committees or official authorities may review the participants' information only when necessary. At the end of the study, the study results may be published in the medical literature, but your identity will not be disclosed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral wisdom teeth in the lower jaw and similar impacted positions
2. Patients with no history of trauma to the head and neck region, no congenital deformities, no degenerative joint disease, patients between the ages of 18 and 25,
3. Patients who have not received any treatment for the adrenal gland in the last 6 months, patients who have not used antidepressant medication in the last 6 months, patients who have no cardiovascular disease, thyroid disease, diabetes, hypertension, renal failure, isolated muscle disease, rheumatological and neurological disease, and patients who have no known psychiatric disorder,
4. Patients with good oral hygiene,
5. Patients who can comply with the scales in the questionnaire form,
6. Patients who have not had surgery on their lower wisdom teeth before,
7. Patients who have not used corticosteroids and anticonvulsant drugs,
8. Patients who have no active caries and pulpal lesions,
9. Patients who can fill out the questionnaire forms on their own. 10) Patients who have not received radiotherapy in the head and neck region and who do not use drugs that may cause MRONJ.

Exclusion Criteria:

1. Patients who had undergone surgical treatment for their wisdom teeth before the study,
2. Patients with serious systemic diseases and those taking medication,
3. Pregnant and breastfeeding women,
4. Individuals using removable dentures,
5. Those receiving psychiatric treatment and those taking medication,

7. Those with a history of heart infarction, 8. Patients using pacemakers, 9. Individuals with epilepsy and neurological disorders, 10. Patients with habits such as alcohol and drug addiction, 11. Patients with advanced periodontitis, 12. Patients undergoing orthodontic treatment and having unstable occlusions, 13. Patients who have received radiotherapy and those taking medications that may cause MRI.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients living in Afyonkarahisar province and applying for extraction of bilaterally impacted wisdom teeth
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | preoperative and postoperative days 2-7
  A 100 mm VAS scale was used to assess postoperative pain. Patients were asked to mark the appropriate part of their pain on the scale during preoperative and postoperative 2nd-7th day controls. In order to standardize analgesic use, patients were informed verbally and in writing that the first analgesic should be taken 1 hour after the operation and then every 8 hours for 3 days, regardless of pain.
Evaluation of Edema | preoperative and postoperative days 2-7
  In the postoperative edema assessment, the tragus, soft tissue pogonion, lateral canthus of the eye, gonion point on the mandible angulus and commissura labiorum were used as anatomical reference points. In the measurements; tragus-lateral canthus, tragus-commissura lobiorum, tragus-soft tissue pogonion, tragus-gonion and gonion-lateral canthus lengths were measured with a flexible ruler and calculated linearly. Preoperative measurement values were accepted as basic values and measurements on postoperative 2nd and 7th days were compared both between the groups and on the preoperative measurement values. Data were created and evaluated by taking the arithmetic average of the measured distances.
Evaluation of Trismus | preoperative and postoperative days 2-7
  The amount of trismus was assessed by measuring the distance between the mesial corners of the right maxillary and mandibular central incisors at maximum mouth opening immediately before the operation and on the 2nd and 7th postoperative days.
Evaluation of Salivary Cortisol | preoperative and postoperative days 2-7
  Before starting the impacted tooth surgery, patients spit into 1.5 ml tubes at 08:30 or 15:30 depending on their groups; 48 hours after surgery and on the 7th day, and these tubes were stored in the refrigerator at -22 degrees. The samples in these tubes were then examined with the 'Human Cor (Cortisol) ELISA Kit- ELK8526' ELISA kits with a measurement sensitivity of 1.02 ng/mL and a measurement range of 3.13-200 ng/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montgomery MT, Hogg JP, Roberts DL, Redding SW. The use of glucocorticosteroids to lessen the inflammatory sequelae following third molar surgery. J Oral Maxillofac Surg. 1990 Feb;48(2):179-87. doi: 10.1016/s0278-2391(10)80207-1. PMID 2405122
- [Background] Chung S, Son GH, Kim K. Circadian rhythm of adrenal glucocorticoid: its regulation and clinical implications. Biochim Biophys Acta. 2011 May;1812(5):581-91. doi: 10.1016/j.bbadis.2011.02.003. Epub 2011 Feb 12. PMID 21320597
- [Background] Balbo M, Leproult R, Van Cauter E. Impact of sleep and its disturbances on hypothalamo-pituitary-adrenal axis activity. Int J Endocrinol. 2010;2010:759234. doi: 10.1155/2010/759234. Epub 2010 Jun 9. PMID 20628523